CLINICAL TRIAL: NCT00510263
Title: A Multicentre Placebo-Controlled Evaluation of Prednisolone and/or Valaciclovir for the Treatment of Bell's Palsy
Brief Title: Scandinavian Bell's Palsy Study
Acronym: SBPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: GlaxoSmithKline (Industry); Pfizer (Industry)
Responsible Party: Mats Engström, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 151:1828/99
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Bell's Palsy
Keywords: Prednisolone; Valacyclovir
MeSH Terms: conditions — Bell Palsy | interventions — Prednisolone; Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Prednisolone + placebo
- 2 (Experimental)
  Interventions: Drug: Valaciclovir + placebo
- 3 (Experimental)
  Interventions: Drug: Prednisolone + valaciclovir
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo + placebo

INTERVENTIONS:
Drug: Prednisolone + placebo — Prednisolone 5 mg 12 tablets per day for 5 days, tapering 2 tablets per day until day 10. Placebo 2 tablets 3 times daily for 7 days.
  Arms: 1
Drug: Valaciclovir + placebo — Valaciclovir 500 mg 2 tablets 3 times daily for 7 days. Placebo tablets 12 per day for 5 days, tapering 2 tablets per day until day 10.
  Arms: 2
Drug: Prednisolone + valaciclovir — Prednisolone 5 mg 12 tablets per day for 5 days, tapering 2 tablets per day until day 10. Valaciclovir 500 mg 2 tablets 3 times daily for 7 days.
  Arms: 3
Drug: Placebo + placebo — Placebo 5 mg 12 tablets per day for 5 days, tapering 2 tablets per day until day 10. Placebo 2 tablets 3 times daily for 7 days.
  Arms: 4

SUMMARY:
The main objective of this study is to study the effects of prednisolone and valaciclovir, with equal importance, compared to placebo for the treatment of Bell´s palsy. The combination of prednisolone and valaciclovir will also be studied.

DETAILED DESCRIPTION:
Study Design:

This is a multicentre randomised double-blind placebo-controlled study.

Study medication:

Prednisolone 60 mg per day for 5 days, after that tapering 10 mg per day for a total treatment time of 10 days. Valaciclovir 1000 mg 3 times per day for 7 days. Prednisolone and valaciclovir are used in combination or separately. One patient of four receives placebo.

Study Duration:

Study medication will be taken during 10 days. The subjects will be followed for 12 months after initiation of treatment. Follow-up visits will be 11-15 days after start of therapy and at 1, 2, 3, 6 and 12 months after the onset of palsy.

Study Setting:

The study will be conducted in 17 ENT-clinics in Sweden and Finland, which will be monitored by the members of the board of the Scandinavian Bells Palsy Study (SBPS)

Study Subjects:

Otherwise healthy subjects with unilateral acute idiopathic facial palsy. A total of 800 subjects will be included in the study.

Study Treatments:

The subjects will be randomised to one of the following treatment arms for oral administration of study drug:

1. Prednisolone + placebo
2. Valaciclovir + placebo
3. Prednisolone + valaciclovir
4. Placebo + placebo

Treatment will be initiated within 72 hours of onset of palsy and continued during 10 days.

Measurements:

The first follow-up clinical examination is scheduled within 3 days after completed treatment. Further follow-up visits are scheduled at 1, 2, 3 and 6 months from onset of palsy. If complete recovery has occurred at the 2 month visit, the 3 and 6 months visits are not necessary. If complete recovery is present at 3 months the 6 month visit can be excluded. A final follow-up exam is always performed at 12 months. The clinical examination includes a routine examination of ear, nose and throat, grading of the palsy according to the Sunnybrook and House Brackmann grading scales and registration of other symptoms as pain, eye irritation, dysacusis and impaired taste. Blood tests for Lyme Borreliosis are drawn at the acute (the first) visit and at the follow-up visit at 2 months.

Primary Endpoint:

The primary endpoint will be the time to complete clinical recovery (defined as 100 on the Sunnybrook facial nerve grading scale) from Bell's palsy. The subjects will be categorised as healed or not healed at months 1, 2, 3, 6 or 12 months. Treatments will be compared using the Generalized Wilcoxon rank sum test. Patients where data are missing and there is no healing time will be included as censored at the last visit when the patient was not healed.

Secondary endpoints:

The secondary endpoints of this study are comparisons between the different treatment arms with regard to:

* Proportion of patients with complete healing of palsy compared to those with incomplete healing at12 months after onset.
* Influence on outcome at 12 months by time in hours from onset of palsy until beginning of study medication.
* Proportion of patients that develop severe palsy during the first week from onset.
* The total duration of pain, in or around the ipsilateral ear or the ipsilateral side of the face, from onset of palsy.
* The proportion of subjects with severe pain (more than VAS 3) in the different treatment arms.
* Occurrence of synkinesia in the different treatment arms at any time.
* Occurrence of facial spasm or contracture in the different treatment arms at any time.
* Severity of remaining facial symptoms in patients not healed at 12 months and at each prescheduled study visit as recorded by Sunnybrook Facial Grading System.

Safety Evaluations:

Adverse events will be assessed during the first study month. Adverse events will be reported in the patient's files and in the patient CRF for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Be in good general health and between 18 and 75 years of age.
2. Have an acute peripheral unilateral idiopathic facial palsy.
3. Not more than 72 hours must have passed after onset of palsy before initiating study medication.
4. The subjects must provide their freely given written informed consent.

Exclusion Criteria:

1. Subjects who have used any antiherpetic medication, except locally applied formulations, within the last 2 weeks.
2. Subjects with ongoing systemic steroid medication for another disease.
3. Pregnant women or nursing mothers.
4. Subjects with diabetes.
5. Subjects presently suffering from gastric or duodenal ulcers. If there is a history of previous peptic ulcers or dyspepsia prophylactic medication must be prescribed and taken during study.
6. Subjects with a history of tuberculosis.
7. Subjects with psychiatric diagnosis that are at risk to be influenced by the study drugs or that might affect the patient´s ability to complete this study.
8. Subjects with a hypertension not well controlled.
9. Subjects with a present, or a history of, serious heart disease.
10. Subjects with a history of glaucoma.
11. Subjects with a history of hepatic disease.
12. Subjects with other neurological diseases.
13. Subjects with a history of renal diseases or a known creatinine clearance of < 30mL/min.
14. Subjects with acute otitis or a history of ipsilateral chronic otitis.
15. Subjects with a history of recent head injury.
16. Fertile, sexually active women not employing acceptable methods of contraception and/or women planning to become pregnant during the period with intake of study medication.
17. Subjects with a history of immunodeficiency syndromes.
18. Subjects with an allergy or sensitivity to aciclovir or valaciclovir, famciclovir or ganciclovir.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2001-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the time to complete clinical recovery from Bell's palsy. | 1, 2, 3, 6 or 12 months.

SECONDARY OUTCOMES:
Proportion of patients with complete healing of palsy compared to those with incomplete healing at 12 months after onset. | 12 months
Influence on outcome at 12 months by time in hours from onset of palsy until beginning of study medication. | 12 months
Proportion of patients that develop severe palsy during the first week from onset. | One week
The total duration of pain, in or around the ipsilateral ear or the ipsilateral side of the face, from onset of palsy. | Two months
The proportion of subjects with severe pain (more than VAS 3) in the different treatment arms. | Two months
Occurrence of synkinesia in the different treatment arms at any time. | 12 months
Occurrence of facial spasm or contracture in the different treatment arms at any time. | 12 months
Severity of remaining facial symptoms in patients not healed at 12 months and at each prescheduled study visit. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mats Engstrom, M.D., Ph.D., Principal Investigator — Uppsala University, Sweden; Lars Jonsson, M.D., Ph.D., Study Director — Uppsala University, Sweden

REFERENCES:
- [Derived] Berg T, Bylund N, Marsk E, Jonsson L, Kanerva M, Hultcrantz M, Engstrom M. The effect of prednisolone on sequelae in Bell's palsy. Arch Otolaryngol Head Neck Surg. 2012 May;138(5):445-9. doi: 10.1001/archoto.2012.513. PMID 22652942
- [Derived] Engstrom M, Berg T, Stjernquist-Desatnik A, Axelsson S, Pitkaranta A, Hultcrantz M, Kanerva M, Hanner P, Jonsson L. Prednisolone and valaciclovir in Bell's palsy: a randomised, double-blind, placebo-controlled, multicentre trial. Lancet Neurol. 2008 Nov;7(11):993-1000. doi: 10.1016/S1474-4422(08)70221-7. Epub 2008 Oct 10. PMID 18849193